CLINICAL TRIAL: NCT00222807
Title: Schizophrenia, Antipsychotic Treatment and the Risk for Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: American Association for Geriatric Psychiatry (Other); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 0306110
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2016-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Delusional Disorder
Keywords: schizophrenia, psychosis, type 2 diabetes mellitus
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples are collected, stored at minus 70 degree C and analyzed in batches.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This preliminary study aims to investigate the mechanism of higher rates of type 2 diabetes mellitus in patients with schizophrenia. As part of the study, we collect neuroendocrine-immune data on patients with first episode, treatment naive psychosis, patients with newly diagnosed schizophrenia and normal healthy controls.

Regardless the treatment status, we collect the same neuroendocrine-immune data on the participants after 2 months.

DETAILED DESCRIPTION:
This preliminary study aims to investigate the mechanism of higher rates of type 2 diabetes mellitus in patients with schizophrenia. As part of the study, we collect neuroendocrine-immune data on patients with first episode, treatment naive psychosis, patients with newly diagnosed schizophrenia and normal healthy controls.

Regardless the treatment status, we collect the same neuroendocrine-immune on the participants (patients and controls) after 2 months. Thus, our study does not control treatment. Patients take treatment in consultation with their physician. Some of them even decide not to take any medications. At the 2nd visit, we do ask them about the the medications they are taking if any.

ELIGIBILITY:
Inclusion Criteria:

* Psychotic disorder as per DSM-IV criteria of the American Psychiatric Association

Exclusion Criteria:

* Diabetes, type 1 or 2
* Prominent substance abuse (i.e. psychotic symptoms attributable entirely to substance use)
* Age above 50 or age below 14

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with psychosis
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2003-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ripu D Jindal, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States